CLINICAL TRIAL: NCT00016159
Title: Phase II Study Of Combined Modality Postremission Therapy As Determined By Molecular Response (Adaptive Regulation) In The Treatment Of Acute Promyelocytic Leukemia (APL)
Brief Title: Chemotherapy Plus Monoclonal Antibody in Treating Patients With Acute Promyelocytic Leukemia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 00-072; MSKCC-00072; NCI-H01-0073
Record Dates: First submitted 2001-05-06; First posted 2003-01-27 (Estimated); Last update posted 2013-01-16 (Estimated); Status verified 2013-01

CONDITIONS: Leukemia
Keywords: adult acute myeloid leukemia in remission; childhood acute myeloid leukemia in remission; adult acute promyelocytic leukemia (M3); childhood acute promyelocytic leukemia (M3); adult acute myeloid leukemia with t(15;17)(q22;q12)
MeSH Terms: conditions — Leukemia; Leukemia, Promyelocytic, Acute | interventions — Filgrastim; lintuzumab; Arsenic Trioxide; Idarubicin; Tretinoin

INTERVENTIONS:
Biological: filgrastim
Biological: lintuzumab
Drug: arsenic trioxide
Drug: idarubicin
Drug: tretinoin

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Monoclonal antibodies can locate tumor cells and either kill them or deliver tumor-killing substances to them without harming normal cells. Combining monoclonal antibody therapy with chemotherapy may kill more cancer cells.

PURPOSE: Phase II trial to study the effectiveness of combination chemotherapy and monoclonal antibody in treating patients who have acute promyelocytic leukemia.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the disease-free and overall survival of patients with acute promyelocytic leukemia in clinical complete remission following tretinoin-based induction therapy treated with monoclonal antibody HuG1-M195, arsenic trioxide, idarubicin, and tretinoin.
* Determine the rate of molecular complete remission in patients treated with this regimen.
* Determine the toxicity of this regimen in this patient population.
* Determine the number and length of hospitalizations of patients treated with this regimen.

OUTLINE: Patients receive monoclonal antibody HuG1-M195 (MOAB HuM195) IV over 40-60 minutes twice weekly for 3 weeks. Approximately 2-4 weeks after completion of MOAB HuM195, patients receive arsenic trioxide IV over 1-4 hours daily for a total of 25 days with no more than 5 days between doses.

Beginning approximately 4-6 weeks after completion of arsenic trioxide, patients receive idarubicin IV daily on days 1-3 or 1-4 and filgrastim (G-CSF) subcutaneously daily beginning on day 5 or 6 and continuing until blood counts recover. Treatment repeats every 4 weeks for patients who remain RT-PCR positive or are newly converted to RT-PCR negative (molecular complete remission) following a prior course of idarubicin for a maximum of 3 courses. Patients who remain RT-PCR positive following course 3 of idarubicin receive no further treatment on study.

Beginning 3 months after completion of idarubicin, patients in molecular complete remission receive oral tretinoin daily for 14 days. Treatment repeats every 3 months for a total of 6 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed monthly.

PROJECTED ACCRUAL: Approximately 35 patients will be accrued for this study within 2-3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of acute promyelocytic leukemia by positive RT-PCR assay for PML/RAR-alfa rearrangement or a t(15;17) karyotype

  * Achieved clinical complete remission within the past 1-2 months
  * Prior induction therapy must have contained tretinoin
* No other acute myeloid leukemia diagnosis

PATIENT CHARACTERISTICS:

Age:

* Any age

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* Bilirubin less than 2 mg/dL
* Transaminases no greater than 3 times upper limit of normal

Renal:

* Creatinine less than 2 mg/dL OR
* Creatinine clearance greater than 60 mL/min

Cardiovascular:

* Ejection fraction normal or greater than 50% by echocardiogram or MUGA

Other:

* No other concurrent active malignancy
* No other serious or life-threatening condition that would preclude study
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for at least 4 months after study

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* See Disease Characteristics
* At least 1 week since prior retinoids

Endocrine therapy:

* Not specified

Radiotherapy:

* Not specified

Surgery:

* Not specified

Other:

* No prior postremission therapy of any form

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2000-11; Primary Completion 2007-03 (Actual)

PRIMARY OUTCOMES:
reverse transcriptase-polymerase chain reaction negativity

CONTACTS AND LOCATIONS:
Overall Officials: Joseph G. Jurcic, MD, Study Chair — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States